CLINICAL TRIAL: NCT01025245
Title: Effect of Intraoperative Magnesium on Remifentanil-induced Postoperative Hyperalgesia After Thyroidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Yuen Hee Shim / Associate professor of Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Reseach Institute, Yonsei University College of Medicine, Seoul, Republic of Korea
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2009-0511
Record Dates: First submitted 2009-11-27; First posted 2009-12-03 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Hyperalgesia
Keywords: Remifentanil induced postoperative hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- remifentanil, MgSO4 (Experimental): Experimental 1 : Intraoperative remifentanil infusion at 0.2 ㎍/㎏/min and MgSO4 30 mg/kg IV at the induction followed by intraoperative infusion at 10 mg/kg/hr Drug : remifentanil, MgSO4 Experimental 2 : Intraoperative remifentanil infusion at 0.2 ㎍/㎏/min and normal saline Drug : remifentanil Active comparator : Intraoperative remifentanil infusion at 0.05 ㎍/㎏/min and normal saline Drug : remifentanil
  Interventions: Drug: remifentanil, MgSO4

INTERVENTIONS:
Drug: remifentanil, MgSO4 — Patients undergoing thyroidectomy will be randomly assigned to one of three groups. Remifentanil will be infused intraoperatively at 0.05 ㎍/㎏/min (group Ⅰ) or 0.2 ㎍/㎏/min (group Ⅱ & Ⅲ). Patients in group Ⅲ will be received 30 ㎎/㎏ MgSO4 at the induction of general anesthesia followed by a maintenance infusion of 10 ㎎/㎏/hr intraoperatively until skin closure.

SUMMARY:
The purpose of this study is to study the effect of intraoperative magnesium on remifentanil-induced postoperative hyperalgesia after thyroidectomy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thyroidectomy,
* Age 20-65,
* American Society of Anesthesiologists physical status classification I or II.

Exclusion Criteria:

* History of chronic pain, Regular use of analgesic, antiepileptic or antidepressive drugs,
* History of drug & alcohol abuse,
* Psychiatric disorder,
* Use of opioids within 24hrs,
* Renal disease with decreased GFR,
* Neuromuscular disease, Severe cardiac disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Tactile pain thresholds adjacent to the surgical wound assessed by von Frey hair before the induction and at postoperative 24 & 48 hrs | postoperative 48 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea